CLINICAL TRIAL: NCT01060631
Title: "Assessment of the Influence of Intracranial Space Occupying Lesions on the Reliability Off Monitoring of the Bispectral Index for Detection of Return of Consciousness."
Brief Title: Influence of Intracranial Lesions on Bispectral Index
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Dr. U. Beese, Department of Anaesthesiology, University Medical Center Groningen,University of Groningen
Other Study IDs: BIS001
Record Dates: First submitted 2010-02-01; First posted 2010-02-02 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2009-11

CONDITIONS: Supratentorial Brain Tumor
Keywords: bispectral index; lesions; consciousness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients with frontal or frontotemporal brain tumor.
  Interventions: Device: BIS values at return of consciousness in patients + predicted and measured propofol plasma concentrations
- patients without supratentorial brain tumor.
  Interventions: Device: BIS values at return of consciousness in patients + predicted and measured propofol plasma concentrations

INTERVENTIONS:
Device: BIS values at return of consciousness in patients + predicted and measured propofol plasma concentrations — Difference between left- and rightsided BIS values in patients with supratentorial brain tumor during course and Comparison between predicted and measured propofol plasma concentrations during course of the study
  Groups: patients with frontal or frontotemporal brain tumor.
Device: BIS values at return of consciousness in patients + predicted and measured propofol plasma concentrations — Difference between left- and rightsided BIS values in patients with supratentorial brain tumor during course and Comparison between predicted and measured propofol plasma concentrations during course of the study
  Groups: patients without supratentorial brain tumor.

SUMMARY:
The purpose of this study is to assess whether BIS values at return of consciousness are different in patients with or without brain tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective craniotomy for removal of frontal or frontotemporal brain tumors.
* Control group: Neurosurgical patients without intracranial pathology.

Exclusion Criteria:

* Patient refusal
* Significantly increased intracranial pressure
* Uncontrolled arterial hypertension
* Significant coronary artery disease
* Anticipated difficult airway
* Decreased level of consciousness
* Existing motor weakness dominant arm/hand
* Impaired hearing
* Nausea, vomiting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bilateral BIS values at return of consciousness in patients with and without supratentorial brain tumor.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Bilateral BIS values at return of consciousness in patients with and without supratentorial brain tumor. | one year

SECONDARY OUTCOMES:
Difference between left- and rightsided BIS values in patients with supratentorial brain tumor during course and Comparison between predicted and measured propofol plasma concentrations during course of the study | one year

CONTACTS AND LOCATIONS:
Overall Officials: U Beese, Dr, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Derived] Sahinovic MM, Eleveld DJ, Miyabe-Nishiwaki T, Struys MMRF, Absalom AR. Pharmacokinetics and pharmacodynamics of propofol: changes in patients with frontal brain tumours. Br J Anaesth. 2017 Jun 1;118(6):901-909. doi: 10.1093/bja/aex134. PMID 28549082